CLINICAL TRIAL: NCT02379338
Title: Phase I Pilot Study of Biodistribution, Metabolism and Excretion of Novel Radiotracer [18F]Fluotriopride ([18F]FTP) by PET/CT
Brief Title: Study of Radiotracer [18F]Fluortriopride ([18F]FTP) by PET/CT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 820959
Record Dates: First submitted 2015-02-12; First posted 2015-03-04 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Dopamine D3 receptor
MeSH Terms: interventions — 16-fluoro-4-thiapalmitic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynamic Brain Cohort (Experimental): The Dynamic Brain cohort will include up to 10 patients who will undergo a dynamic brain [18F]Fluortriopride PET/CT scan over a period of approximately 2 hours. Subjects in this cohort will also undergo a research brain MRI, generally on a separate day from the PET/CT.
  Interventions: Drug: [18F]Fluortriopride
- Biodistribution Cohort (Experimental): The Biodistribution cohort will include up to10 patients who will undergo a series of whole body biodistribution [18F]Fluortriopride PET/CT scans over a period of approximately 4 hours.
  Interventions: Drug: [18F]Fluortriopride

INTERVENTIONS:
Drug: [18F]Fluortriopride — All subjects will receive a [18F]Fluortriopride PET/CT scan
  Other Names: [18F]FTP

SUMMARY:
In this phase 1 pilot study, positron emission tomography (PET/CT) imaging will be used to determine the biodistribution, metabolism and excretion of a novel radiotracer [18F]Fluortriopride ([18F]FTP).

DETAILED DESCRIPTION:
[18F]FTP is a novel radioactive tracer that has shown potential in labeling dopamine D3 receptors through PET/CT imaging. This is a phase 1 study design meant to evaluate safety, biodistribution and brain uptake of [18F]FTP in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age
2. "Healthy volunteer" is defined as being in good general health in the opinion of an investigator (controlled diabetes, controlled hypertension or other well controlled chronic medical conditions may be allowed at the discretion of an investigator if they do not believe they will increase patient risk or interfere with the collection of imaging data, specific excluded conditions are described under exclusion criteria)
3. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant at the time of screening will not be eligible for this study, urine or blood pregnancy test will be performed in women of child-bearing potential at screening.
2. Body Mass Index (BMI) > 35
3. Sustained uncontrolled hypertension (Systolic blood pressure greater than 160 mm Hg and/or diastolic blood pressure greater than 110 mm Hg) at screening intake session. If either of the pressure values is above the stated limits on the initial assessment, blood pressure may be re-tested twice after initial assessment at five minute intervals (for a total of 3 blood pressure assessments). The pressure elevation is considered sustained if either the systolic or diastolic pressure values are outside the stated limits for all three assessments, and the subject will be excluded from study participation.
4. History of epilepsy or seizure disorder as assessed by medical record review and/or self-reported
5. History of head trauma, that in the opinion of an investigator may interfere with the uptake of [18F]FTP as assessed by medical record review and/or self-reported
6. History of Post-Traumatic Stress Disorder (PTSD), bipolar disorder, schizophrenia or psychotic disorder as assessed by medical record review and/or self-reported
7. Use of dopaminergic CNS stimulants (prescription, over-the counter or recreational drugs) within 30 days of screening intake visit , as assessed by review of health history form and concomitant medication review at screening intake visit (from medical record and/or self-reported) that are deemed by a physician investigator to have a potential influence on the binding of [18F]FTP
8. Positive urine drug screen at the screening intake visit
9. Self-reported current alcohol consumption that exceeds greater than 25 drinks per week
10. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
11. Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Determine biodistribution of the radioactive investigational drug ([18F]fluortriopride) in healthy volunteers and calculate human dosimetry. | 1 week
  Assessing the biodistribution of the radioactive investigational drug ([18F]fluortriopride) and calculation of human dosimetry in healthy volunteers are completed with MRI results from Dynamic Brain cohort, PET/CT results and laboratory results.
Demonstrate the feasibility of imaging the brain with the dopamine D3 receptor imaging agent [18F]fluortriopride | 1 week
  Participants will complete an anatomical MRI scan on an MRI scanner (without contrast) to enable precise anatomic location of the PET scan results. MRI and PET images will be co-registered so that the anatomical structures observed on the MRI can be accurately outlined on the PET scans for analysis.

SECONDARY OUTCOMES:
Evaluate the safety of [18F]fluortriopride | 24 hours
  Safety of the radioactive investigational drug ([18F]fluortriopride) as measured by the number of participants with adverse events and significant changes in laboratory and/or PET/CT results.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Dubroff, MD, PhD, Principal Investigator — Hospital of University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Mach RH, Tu Z, Xu J, Li S, Jones LA, Taylor M, Luedtke RR, Derdeyn CP, Perlmutter JS, Mintun MA. Endogenous dopamine (DA) competes with the binding of a radiolabeled D(3) receptor partial agonist in vivo: a positron emission tomography study. Synapse. 2011 Aug;65(8):724-32. doi: 10.1002/syn.20891. Epub 2011 Mar 21. PMID 21132811